CLINICAL TRIAL: NCT06922071
Title: The REMINDER4Care Program for Older Adults Supported by Residential and Daycare Facilities
Acronym: REMINDER4Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Principal Investigator, Catarina Baptista, Principal Investigator, University of Coimbra
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: RCTREMINDER4Care
Record Dates: First submitted 2025-03-31; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Dementia Risk Factors; Prevention; Cognitive Health
Keywords: Dementia Risk Factors; Prevention; Health; Aging; Residential and Daycare Facilities; Lifestyle

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- REMINDER4Care intervention (Experimental): In this arm, participants will receive the intervention - REMINDER4Care. REMINDER4Care is a 20-session group program that includes psychoeducation about the brain, social skills training, using cognitive aids, setting personal goals, and practicing mindfulness.
  Interventions: Other: REMINDER4Care
- Waiting-list group (No Intervention): In this arm, participants will be a waiting-list group and receive the REMINDER4Care interventions after the study ends (after the post-interventions).

INTERVENTIONS:
Other: REMINDER4Care — REMINDER4Care was an adapted version of the original REMINDER program, tailored to the characteristics, needs, and interests of older adults in RDF.
  The REMINDER4Care intervention includes 20 face-to-face group sessions, each approximately 60 to 75 minutes, held twice a week over ten weeks. This program aims to optimize memory, attention, executive function, and emotional regulation while promoting lifestyle habits that protect the aging brain. The sessions include brain health education, cognitive exercises, compensatory memory strategies, training for managing personally relevant goals (with goal setting), and stress management techniques (compassion-based therapies, relaxation methods, and mindfulness). Social support and emotion regulation strategies (like attention management, positive cognitive reappraisal, and reframing speech) were included to address psychosocial risk factors like stress, social isolation, and depression.
  Arms: REMINDER4Care intervention

SUMMARY:
Dementia incidence is rising, posing a public health challenge, but 45% of cases can be prevented by addressing modifiable risk factors. Multidomain trials show that lifestyle changes can improve cognitive function and reduce dementia risk (like the FINGER trial). The REMINDER program, a Portuguese-based dementia risk reduction protocol, was developed for community-dwelling older adults aged 55 and above. However, older adults in Residential and Daycare Facilities (RDF) have distinct needs that demand program adaptation to ensure its relevance and effectiveness. In addition, more studies are needed to evaluate the impact of multidomain interventions with older adults in RDF.

To address these challenges, the REMINDER4Care program was developed as a tailored, multidomain intervention to reduce dementia risk. It emphasizes social and cognitive engagement and advances its adaptation and evaluation in Residential and Daycare Facilities (RDF). To assess efficacy, the investigators will perform a Randomized Controlled Trial.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years and older
* RDF users
* Elementary reading and writing skills

Exclusion Criteria:

* Have a clinical diagnosis of dementia and/or Mini-Mental State Examination (MMSE) scores below the cutoff for the presence of dementia (MMSE < 22-27, depending on education level)
* Have a psychiatric or neurological condition that impairs cognition in the long term
* Have sensory and functional deficits that compromise their participation in the neuropsychological assessment and throughout the intervention sessions

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Screening | Screening
  Participants' sociodemographic (e.g., age, marital status, education level) and clinical (presence of medical diagnosis, current medication, sensory issues, mobility deficits, substance use, and hospitalization).
Screening | Screening
  Dementia risk was assessed using the Lifestyle for BRAin health (LIBRA) score, which ranges from -2.1 to 10.6, with higher scores indicating a greater risk of developing dementia.
Cognitive status | Screening and 1-week and 3-months post-intervention
  Global cognition was assessed using Addenbrooke's Cognitive Examination - Revised (ACE-R), a scale with scores ranging from 0 to 100, where higher scores indicate better cognitive functioning.
Mood status | Screening and 1-week and 3-months post-intervention
  Depressive Symptoms: Assessed using the Geriatric Depression Scale (GDS-30), a 30-item scale with scores ranging from 0 to 30, where higher scores indicate greater depressive symptoms.
Cognitive status | Baseline and 1-week and 3-months post-intervention
  Processing Speed: Evaluated with the Symbol Search subtest of the WAIS-III, scored by correct responses within a time limit, with higher scores representing faster processing speed.
Cognitive status | Baseline and 1-week and 3-months post-intervention
  Verbal Initiative: Measured with the Verbal Fluency Test (letters M, R, and alternate category), scored by the number of correct words produced, with higher scores indicating greater verbal initiative.
Perceived social isolation and loneliness | Baseline and 1-week and 3-months post-intervention
  Loneliness: Measured with the UCLA Loneliness Scale (UCLA LS-3), the score was 20 to 80, with higher scores reflecting greater perceived loneliness.
Perceived social network | Baseline and 1-week and 3-months post-intervention
  Social Networks: Evaluated using Lubben's Brief Social Network Scale (LSNS-6), scored from 0 to 30, where higher scores indicate a stronger social network.
Functionality status | Baseline and 1-week and 3-months post-intervention
  Functional abilities: This is measured using the IAFAI (Informant Assessment of Functioning in Aging and Intellectual Disabilities).
Perceived quality of life | Baseline and 1-week and 3-months post-intervention
  Psychological Well-Being: Assessed using the EBEP-R is a short version of the Psychological Well-Being Scale. Higher scores on the EBEP-R indicate better psychological well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Catarina L. B. Baptista, PhD Student, Principal Investigator — University of Coimbra; Ana Rita E. S. Silva, Doctorate, Study Chair — University of Coimbra; Margarida P. Lima, Doctorate, Study Chair — University of Coimbra; Rosa M. Afonso, Doctorate, Study Chair — University of Beira Interior
Locations (1):
- Faculty of Psychology and Education Sciences, Coimbra, Portugal, Portugal

IPD SHARING:
Plan to Share IPD: Undecided
Open science plans will involve sharing IPD with other researchers, clearly anonymized, to promote the study's replication. The investigators are still developing the strategy for data sharing and will update as soon as it is defined.

REFERENCES:
- See also: Website REMINDER — https://www.remindereomeucerebro.pt/